CLINICAL TRIAL: NCT06371820
Title: ESPRESSO (Epidemiology Strengthened by histoPathology Reports in Sweden)
Acronym: ESPRESSO
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jonas Ludvigsson, Professor, Karolinska Institutet
Other Study IDs: 2014/1287-31/4
Record Dates: First submitted 2024-03-27; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Gastrointestinal Diseases
Keywords: cohort; gallbladder; gut; liver; pancreas; population-based; colon; pathology; endoscopy; celiac; inflammatory bowel disease; colitis; esophagus
MeSH Terms: conditions — Gastrointestinal Diseases; Celiac Disease; Inflammatory Bowel Diseases; Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ESPRESSO [The study has no intervention] — This study has no interventions.

SUMMARY:
The ESPRESSO study is a collection of data from all computerised gastrointestinal histopathology reports in Sweden. This allows us to study risk factors for gastrointestinal disease, as well as the prognosis of gastrointestinal disease.

A review of the study has been published here:

https://pubmed.ncbi.nlm.nih.gov/30679926/

DETAILED DESCRIPTION:
The ESPRESSO study constitutes a novel approach to examine the etiology and prognosis of gastrointestinal disease in which histopathology plays a prominent role. Between 2015 and 2017, all pathology departments (n=28) in Sweden were contacted and asked to procure histopathology record data from the gastrointestinal tract (pharynx to anus), liver, gallbladder, and pancreas. For each individual, local histopathology IT personnel retrieved data on personal identity number, date of histopathology, topography (where the biopsy is taken), morphology (biopsy appearance), and where available free text. In total, between 1965 and 2017, histopathology record data were available in 2.1 million unique individuals, but the number of data entries was 6.1 million because more than one biopsy was performed in many of the study participants. Index individuals with histopathology data were matched with up to five controls from the general population. The investigators also identified all first-degree relatives (parents, children, full siblings), and the index individual's first spouse. The total study population consisted of 13.0 million individuals. Data from all the study participants have been linked to Swedish National Healthcare Registers allowing research not only on such aspects as fetal and perinatal conditions and the risk of future gastrointestinal disease but also on the risk of comorbidity and complications (including cancer and death). Furthermore, the ESPRESSO database allows researchers and practitioners to identify diagnoses and disease phenotypes not currently indexed in national registers (including disease precursors). The ESPRESSO database increases the sensitivity and specificity of already-recorded diseases in the national health registers. This paper is an overview of the ESPRESSO database.

ELIGIBILITY:
Inclusion Criteria:

* Any person with a computerised histopathology record from the gastrointestinal tract including the liver, gallbladder and the pancreas.
* Matched controls to any person with the above histopathology record.
* Spouses and first-degree relatives to any of the above.

Exclusion Criteria:

-None

(this is a registry-based study)

Ages: 0 Years to 110 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Males 45.8% Median age at biopsy: 58 years
Sampling Method: Probability Sample
Enrollment: 13000000 (Actual)
Dates: Start 1965-01-01 (Actual); Primary Completion 2043-05-17 (Estimated); Study Completion 2043-05-17 (Estimated)

PRIMARY OUTCOMES:
Incident Mortality [especially rates] | Currently up until 2022
  Record of death in the Swedish Cause of Death Register. Please note: Different sub-projects will have different primary outcomes.

SECONDARY OUTCOMES:
Incident Cancer | Currently up until 2022
  ICD (international classification of diseases) code in the Swedish nationwide cancer register.
Incident Cardiovascular disease | Currently up until 2022
  ICD (international classification of diseases) code in the Swedish nationwide Patient Register, and where appropriate also the Cause of Death Register
Incident Neurological disease | Currently up until 2022
  ICD (international classification of diseases) code in the Swedish nationwide Patient Register, and where appropriate also the Cause of Death Register
Incident Autoimmune diseases | Currently up until 2022
  ICD (international classification of diseases) code in the Swedish nationwide Patient Register, and where appropriate also the Cause of Death Register

OTHER OUTCOMES:
Please note that the recorded outcomes above are examples. Other outcomes may also be studied. | Currently up until 2022
  ICD codes as above

CONTACTS AND LOCATIONS:
Overall Officials: Jonas F Ludvigsson, MD, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers. (such sharing is not consistent with the rules from the Swedish government agency: Statistics Sweden).

REFERENCES:
- [Result] Ludvigsson JF, Lashkariani M. Cohort profile: ESPRESSO (Epidemiology Strengthened by histoPathology Reports in Sweden). Clin Epidemiol. 2019 Jan 14;11:101-114. doi: 10.2147/CLEP.S191914. eCollection 2019. PMID 30679926